CLINICAL TRIAL: NCT06991842
Title: Effect of Phosphoric Acid Etching Duration on the Performance of Direct Resin-Based Composite Restorations in Permanent Anterior Teeth: A Randomized Controlled Single-Center Trial
Brief Title: Effect of Phosphoric Acid Etching Duration on Direct Resin-Based Composite Restorations in Permanent Anterior Teeth
Acronym: ETCH-PRO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Florin Eggmann (Other)
Responsible Party: Sponsor-Investigator, Florin Eggmann, Sponsor-Investigator, Head of Cariology, University Hospital, Basel, Switzerland
Organization: University Hospital, Basel, Switzerland (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ETCH-PRO; 2025-00584 (Other: EKNZ)
Record Dates: First submitted 2025-05-07; First posted 2025-05-28 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-08

CONDITIONS: Dental Restoration, Permanent; Dental Caries (Disorder); Dental Restoration Failure
Keywords: Resin-based composite; Universal adhesive; Class III restoration; Class IV restoration; Phosphoric acid etching; Adhesive dentistry; Anterior tooth restoration; Permanent dental restoration; Dental bonding; Etch-and-rinse technique; Restorative dentistry
MeSH Terms: conditions — Dental Caries | interventions — Dental Restoration, Permanent

STUDY DESIGN:
Intervention Model Description: This is a single-center, two-arm, parallel-group, randomized controlled trial comparing the clinical outcomes of direct resin-based composite restorations in anterior permanent teeth using either a standard phosphoric acid etching (PAE) protocol or a reduced PAE duration protocol. Each participant is allocated to one of the two groups and receives a single intervention type throughout the study period. No crossover is performed, and all restorative procedures follow standardized protocols, differing only in the PAE regimen.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard PAE Protocol Group (Active Comparator): In this arm, participants will receive a Class III or Class IV resin-based composite (RBC) restoration with a standard etch-and-rinse bonding protocol. Phosphoric acid etching (PAE) will be applied to both enamel and dentin for 15-30 seconds and 10-15 seconds, respectively. After etching, a universal adhesive will be applied, followed by the placement of the RBC using a standard layering technique with separately photo-polymerized increments. The final restoration will be polished to ensure proper contour and surface finish.
  Interventions: Procedure: Permanent dental restoration
- Reduced PAE Duration Protocol Group (Experimental): Participants in this arm will receive Class III or Class IV RBC restorations using a reduced PAE duration protocol. Phosphoric acid etching will be applied simultaneously to both enamel and dentin for a brief 10-second period, followed by the application of the universal adhesive and placement of the RBC. Similar to the standard protocol group, the restoration will be placed using a layering technique with photo-polymerized increments and polished to completion. This group aims to evaluate the effect of a reduced etching time on restorative outcomes compared to the standard PAE protocol.
  Interventions: Procedure: Permanent dental restoration

INTERVENTIONS:
Procedure: Permanent dental restoration — In both study arms, permanent dental restorations are made with resin-based composite in permanent anterior teeth. Both study arms will use identical materials for the resin-based composite restoration (Tetric Plus Flow and Tetric Plus Fill) and universal adhesive (Adhese Universal), with the only difference being the duration of the phosphoric acid etching step. All other aspects of the restorative procedure, such as isolation of the operative field, application techniques, and final polishing, will remain consistent across both arms.

SUMMARY:
The goal of this clinical trial is to learn if reducing the phosphoric acid etching (PAE) time affects the performance of direct resin-based composite (RBC) restorations in permanent anterior teeth. It will also learn about the safety of using a shortened PAE protocol. The main questions it aims to answer are:

Does a shorter PAE time lead to more or less marginal staining in restored teeth?

What sensitivity or other clinical issues do participants experience after restoration using different PAE times?

Researchers will compare a reduced PAE protocol to a standard PAE protocol to see how each affects the outcome of Class III and IV anterior restorations.

Participants will:

Receive one or two direct RBC restorations using either a shortened or standard PAE protocol

Visit the clinic for follow-ups at baseline, and at 1, 2, 3, and 5 years after restoration

Have sensitivity and restoration quality evaluated using clinical exams, photographs, and questionnaires

DETAILED DESCRIPTION:
This clinical trial, "Effect of Phosphoric Acid Etching Duration on the Performance of Direct Resin-Based Composite Restorations in Permanent Anterior Teeth: A Randomized Controlled Single-Center Trial," or ETCH-PRO for short, aims to investigate whether reducing the duration of phosphoric acid etching (PAE) impacts the effectiveness and safety of direct resin-based composite (RBC) restorations in permanent anterior teeth.

Specifically, it seeks to answer:

DOES A SHORTER PAE TIME AFFECT MARGINAL STAINING IN RESTORED TEETH?

WHAT POSTOPERATIVE SENSITIVITY OR OTHER CLINICAL ISSUES DO PARTICIPANTS EXPERIENCE WITH DIFFERENT PAE TIMES?

Researchers at the University Center for Dental Medicine Basel UZB will compare a reduced PAE protocol to a standard PAE protocol. Participants will receive one or two direct RBC restorations using either protocol and attend follow-up visits at baseline (7-10 days post-op), and at 1, 2, 3, and 5 years after restoration. During these visits, sensitivity and restoration quality will be assessed through clinical exams, photographs, and questionnaires.

DETAILED DESCRIPTION

BACKGROUND AND RATIONALE

Phosphoric acid etching (PAE) is crucial for enhancing enamel bond strength in restorative dentistry. When using etch-and-rinse adhesives, PAE is necessary for successful dentin bonding. However, with self-etch adhesives, PAE of dentin is not recommended due to potential negative effects on adhesion.

The increasing use of universal adhesives offers clinicians flexibility in choosing between etch-and-rinse and selective enamel etching techniques. A key challenge with selective enamel etching is the risk of inadvertently etching the dentin, which can compromise adhesion and the longevity of the restoration.

Recent laboratory studies suggest that shortening PAE duration does not negatively affect bond strength, potentially mitigating the risks associated with accidental dentin etching. However, clinical data on the long-term outcomes of direct RBC restorations in anterior teeth using reduced PAE times is limited.

This study aims to address this gap by evaluating the clinical performance of RBC restorations in anterior permanent teeth using a reduced PAE protocol compared to a standard protocol.

The study specifically includes teeth requiring Class III or Class IV restorations due to:

Proximal carious lesions with cavitation

Replacement of defective restorations

Necessary proximal reshaping (e.g., for developmental anomalies, proximal gaps, or esthetic concerns like black triangles)

Class IV cases are strictly limited to non-fracture-related reshaping.

The study operates under the null hypothesis, stating there is no significant difference in clinical outcomes between the two PAE protocols. Confirmation of this could support adopting reduced PAE durations in routine practice, potentially improving procedural efficiency and minimizing iatrogenic effects.

RISK/BENEFIT ASSESSMENT

STUDY OVERVIEW

All procedures adhere to established, evidence-based restorative practices, using CE-marked materials and standardized protocols to ensure patient safety and consistency. This study is classified as Risk Category A according to ClinO, Art. 61, indicating minimal risks and burdens.

ANTICIPATED CLINICAL BENEFITS

While participants may not experience immediate personal benefits, their involvement will contribute valuable data to improve clinical protocols and outcomes for future patients.

RESIDUAL RISKS AND ADVERSE DEVICE EFFECTS (ADES)

The materials used comply with CE marking requirements, presenting minimal residual risks. Minor postoperative discomfort or sensitivity may occur but are considered rare and manageable.

RISKS DUE TO CONCOMITANT TREATMENTS

No specific risks from concomitant treatments are anticipated. Each participant's medical history will be reviewed during screening to monitor potential interactions.

PARTICIPATION RISKS AND SAFETY MEASURES

Participants are fully informed about the study's procedures, potential risks, and the lack of direct benefits. Written informed consent is obtained before participation. Close monitoring will ensure adverse events are promptly addressed.

RISK-MITIGATION STRATEGIES

Comprehensive risk analysis and procedural safeguards

Proper training and calibration of all clinical personnel

Clear patient communication and continuous monitoring

Standardized procedures to minimize discomfort and risks

RISK-BENEFIT ASSESSMENT

The minimal and manageable risks are outweighed by the potential benefits of improving long-term restorative outcomes and informing future best practices.

OBJECTIVES

PRIMARY OBJECTIVE

To compare the frequency of marginal staining in anterior direct RBC restorations between the standard and reduced PAE protocol groups.

SECONDARY OBJECTIVES

To assess the frequency of postoperative hypersensitivity levels following restoration

To comprehensively evaluate the overall quality of the restorations based on clinical, esthetic, and functional parameters

ENDPOINTS

PRIMARY ENDPOINT

Frequency of marginal staining in direct RBC restorations, assessed using the Category A2 guideline from the FDI criteria, incorporating the SQUACE method.

SECONDARY ENDPOINTS

Frequency and severity of pulpal hypersensitivity and pulpal status at 7-10 days post-treatment (FDI criteria B3)

Comprehensive evaluation of restoration quality based on FDI criteria:

Surface luster and surface texture (FDI A1)

Color match (FDI A3)

Caries at the restoration margin (FDI B1)

Dental hard tissue defects (FDI B2)

Fracture of material and retention (FDI F1)

Marginal adaptation (FDI F2)

Proximal contact quality (FDI F3), supplemented by testing with metal matrices (25-100 µm)

Form and contour (FDI F4)

Occlusion and wear (FDI F5)

Patient satisfaction (FDI M1) using a VAS scale (0-10)

Evaluations will be conducted at baseline, 1, 2, 3, and 5 years post-placement. Magnifying loupes and predefined-tip probes (250 µm) will be used. For FDI criteria F2, B1, and B2, margins will be analyzed via the SQUACE method.

STUDY DESIGN

This is a single-center, randomized, controlled trial with two parallel study arms, conducted at the University Center for Dental Medicine Basel UZB.

BLINDING: Assessors and participants are blinded; operators are not, due to procedural differences

COMPARATOR: Conventional etch-and-rinse vs. reduced PAE protocol

ALLOCATION RATIO: 1:1

FRAMEWORK: Non-inferiority design

ELIGIBILITY CRITERIA

INCLUSION CRITERIA

Adults (≥18 years) with signed informed consent

Indication for Class III or IV RBC restoration due to:

Proximal carious lesion with cavitation

Defective restoration requiring replacement

Necessary proximal reshaping

Vital teeth with normal sensitivity

VAS <3 for preoperative sensitivity/biting discomfort

Good oral hygiene and clinical periodontal health

EXCLUSION CRITERIA

Inability to achieve proper isolation

Class IV restorations due to trauma or extensive wear

Missing antagonist tooth without replacement

Intent to bleach within 5 years post-restoration

Allergies to materials used

Pregnancy or lactation

Health conditions impairing participation

SEX AND GENDER CONSIDERATIONS

Sex and gender are not considered significant variables, as restorative needs and outcomes do not vary by these factors. Key influencers include caries risk and technique.

SAMPLE SIZE AND RATIONALE

Total: 66 participants (33 per arm). The size accounts for a 10% dropout rate, with power calculations based on published marginal discoloration data.

STUDY INTERVENTION

All participants receive direct RBC restorations:

TEST GROUP: 10-second total-etch with simultaneous enamel and dentin application

CONTROL GROUP: Standard etch-and-rinse: 15-30 seconds on enamel, 10-15 on dentin

Same materials for both:

Adhesive: Adhese Universal

RBC: Tetric plus Flow and Fill

All procedures follow standardized restorative protocols.

STUDY PROCEDURES

One or two restorations per participant

Recruitment from UZB patient base

Randomization: Computer-generated (Castor), stratified by age, gender, and restoration class

Assessments:

FDI criteria (blinded evaluator)

VAS for sensitivity

Intraoral photos at all timepoints

FOLLOW-UP SCHEDULE:

Baseline (7-10 days post-op)

1, 2, 3, and 5 years

STUDY DURATION AND SCHEDULE

Total duration: ~6 years

First subject in: May 2025

Last subject out: May 2031

STUDY CENTER

University Center for Dental Medicine Basel UZB Department of Periodontology, Endodontology, and Cariology Mattenstrasse 40 CH-4058 Basel, Switzerland

STATISTICAL CONSIDERATIONS

Significance level (α): 0.05

Power (1-β): 0.80

Kaplan-Meier survival analysis and log-rank test for group comparison

DATA PRIVACY

Compliance with ISO 14155, GDPR, HIPAA

Data pseudonymized and securely stored (Castor)

Access restricted to authorized personnel

Lay summary results shared with participants

Data archived for 20 years

ETHICAL CONSIDERATIONS

Routine, low-risk intervention

Excludes vulnerable populations

Equal gender representation ensured

Minimal risks, mitigated through staff training and close monitoring

Aim: Advance restorative dentistry and improve long-term patient outcomes

ELIGIBILITY:
Inclusion Criteria:

Signed informed consent by the participant

Age 18 years or older

Indication for a Class III or Class IV resin-based composite (RBC) restoration on an anterior permanent tooth due to one or more of the following conditions:

Proximal carious lesion with cavitation

Defective restoration requiring replacement

Necessary proximal reshaping due to developmental anomalies (e.g., peg teeth, proximal gaps from Bolton discrepancies, orthodontic tooth position, or esthetic concerns like black triangles caused by periodontal tissue recession)

Vital teeth with regular sensitivity

Sufficient language skills to understand and comply with study procedures

Preoperative Visual Analog Scale (VAS) scores < 3 for tooth sensitivity and biting discomfort

Good oral hygiene, including the ability to maintain effective oral hygiene

Clinical periodontal health (intact periodontium or a reduced periodontium due to non-periodontal causes or after periodontal treatment)

Exclusion Criteria:

Inability to achieve sufficient isolation and contamination control during restorative procedures

Class IV restoration required due to crown fracture, crown-root fracture, extensive tooth wear, or carious lesion affecting the incisal edge

Missing antagonist tooth without prosthodontic replacement

Intent to undergo professional tooth bleaching within five years following the Class III or IV restoration (Note: Professional tooth bleaching must be completed at least two weeks prior to study enrollment)

Known or suspected allergy to any constituents of the materials used (e.g., methacrylates or local anesthetics)

Pregnancy or lactation

Acute or chronic health conditions that may impair study participation (e.g., systemic diseases, oral conditions, or treatments that interfere with study procedures)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2031-05-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Frequency of Marginal Staining in Direct Resin-Based Composite Restorations of Anterior Teeth | Baseline, 1, 2, 3, and 5 years post-restoration placement
  The primary outcome measure is the frequency of marginal staining in direct resin-based composite restorations placed in anterior permanent teeth, assessed at baseline and at 1, 2, 3, and 5 years post-restoration. Marginal staining will be evaluated using the Category A2 guideline from the FDI criteria. This outcome aims to determine if the duration of phosphoric acid etching affects the incidence of marginal staining over time.

SECONDARY OUTCOMES:
Postoperative Sensitivity/Pulpal Status | 7-10 days post-restoration placement
  Postoperative sensitivity will be assessed according to the FDI category B3 criterium.
Fracture of material/retention | Baseline, 1, 2, 3, and 5 years post-restoration placement
  Fracture of material/retention will be assessed according to the FDI criterium F1.
Marginal adaptation | Baseline, 1, 2, 3, and 5 years post-restoration placement
  Marginal adaptation will be assessed according to the FDI criterium F2.
Proximal contact point | Baseline, 1, 2, 3, and 5 years post-restoration placement
  Proximal contact point will be assessed according to the FDI criterium F3.
Form/contour | Baseline, 1, 2, 3, and 5 years post-restoration placement
  Form/contour will be assessed according to the FDI criterium F4.
Occlusion/wear | Baseline, 1, 2, 3, and 5 years post-restoration placement
  Occlusion/wear will be assessed according to the FDI criterium F5.
Caries at restoration margins | Baseline, 1, 2, 3, and 5 years post-restoration placement
  Caries at restoration margins will be assessed according to the FDI criterium B1.
Dental hard tissue defects at the restoration margin | Baseline, 1, 2, 3, and 5 years post-restoration placement
  Dental hard tissue defects at the restoration margin will be assessed according to the FDI criterium B2.
Surface luster/surface texture | Baseline, 1, 2, 3, and 5 years post-restoration placement
  Surface luster/surface texture will be assessed according to the FDI criterium A1.
Color match | Baseline, 1, 2, 3, and 5 years post-restoration placement
  Color match will be assessed according to the FDI criterium A3.
Patient's view | Baseline, 1, 2, 3, and 5 years post-restoration placement
  Patient's view will be assessed according to the FDI criterium M1.

CONTACTS AND LOCATIONS:
Overall Officials: Florin Eggmann, PD Dr. med. dent., Principal Investigator — University of Basel
Locations (1):
- University Center for Dental Medicine Basel UZB, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided
Plan Description A decision has not yet been made regarding the sharing of individual participant data (IPD) collected in this study. Factors under review include participant consent, data privacy protections, institutional policies, and applicable regulations. If IPD sharing is determined to be appropriate, the data will be de-identified and made available to qualified researchers through a secure platform, in accordance with relevant ethical and legal standards. This record will be updated with access details if and when data sharing becomes available.
  Access Criteria If IPD becomes available for sharing, access will be granted to qualified researchers upon request, subject to approval of a data use agreement and verification of compliance with ethical and legal standards.

REFERENCES:
- [Background] Wong J, Tsujimoto A, Fischer NG, Baruth AG, Barkmeier WW, Johnson EA, Samuel SM, Takamizawa T, Latta MA, Miyazaki M. Enamel Etching for Universal Adhesives: Examination of Enamel Etching Protocols for Optimization of Bonding Effectiveness. Oper Dent. 2020 Jan/Feb;45(1):80-91. doi: 10.2341/18-275-L. Epub 2019 Jun 21. PMID 31226005
- [Background] Tsujimoto A, Fischer N, Barkmeier W, Baruth A, Takamizawa T, Latta M, Miyazaki M. Effect of Reduced Phosphoric Acid Pre-etching Times on Enamel Surface Characteristics and Shear Fatigue Strength Using Universal Adhesives. J Adhes Dent. 2017;19(3):267-275. doi: 10.3290/j.jad.a38437. PMID 28597008
- [Background] Burrer P, Dang H, Par M, Attin T, Taubock TT. Effect of Over-Etching and Prolonged Application Time of a Universal Adhesive on Dentin Bond Strength. Polymers (Basel). 2020 Dec 3;12(12):2902. doi: 10.3390/polym12122902. PMID 33287394
- [Background] Amran T, Meier D, Amato J, Connert T, Blatz MB, Weiger R, Eggmann F. Accuracy of Selective Enamel Etching: A Computer-assisted Imaging Analysis. Oper Dent. 2023 Sep 1;48(5):538-545. doi: 10.2341/22-114-L. PMID 37635464

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-04-22): https://cdn.clinicaltrials.gov/large-docs/42/NCT06991842/Prot_SAP_000.pdf
  • Informed Consent Form (2025-04-19): https://cdn.clinicaltrials.gov/large-docs/42/NCT06991842/ICF_001.pdf